CLINICAL TRIAL: NCT06514833
Title: Effects of Regular Napping in Pregnant Women With Sleep Disturbances on Offspring Neurodevelopment
Brief Title: Effects of Napping in Pregnant Women With Sleep Disturbances on Offspring Neurodevelopment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: XH-24-006
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Sleep
Keywords: Sleep disturbance; Neurodevelopment
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors responsible for conducting the neurodevelopment tests are blinded to the group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nap (Experimental): The experimental group will receive lifestyle recommendations to nap regularly
  Interventions: Behavioral: lifestyle recommendations to nap regularly
- No nap (Other): The control group would not receive lifestyle recommendations to nap regularly
  Interventions: Other: No recommendations to nap regularly

INTERVENTIONS:
Behavioral: lifestyle recommendations to nap regularly — Participants will receive lifestyle recommendations to nap regularly for 15-30 minutes between 12:00 and 15:00
  Arms: Nap
Other: No recommendations to nap regularly — No lifestyle recommendations to nap regularly
  Arms: No nap

SUMMARY:
To examine the effects of napping in pregnant women with sleep disturbances on offspring neurodevelopment, the researchers will recruit 80 pregnant women with sleep disturbances. These women will receive lifestyle recommendations to nap regularly and will choose whether or not to nap. The participants will wear wrist-worn accelerometers to record their 24-hour sleep patterns for seven consecutive days during the early, middle, and late stages of pregnancy. The neurodevelopment of their offspring will be assessed at 6 months, 12 months, 18 months, and 2 years of age.

DETAILED DESCRIPTION:
Participants will be recruited based on the Early Life Plan Project, an ongoing hospital-based prospective birth cohort study. Pregnant women will be recruited at the time of booking for prenatal care. The sleep patterns of pregnant women will be assessed at 12-16 weeks of gestation using the Pittsburgh Sleep Quality Index (PSQI) questionnaire. Women with a PSQI score greater than 5 and who self-report as not being habitual nappers in the last 3 months will be recruited. These women will receive lifestyle recommendations to nap regularly for 15-30 minutes between 12:00 and 15:00. Whether they adopt this lifestyle change or the actual duration of their naps will be entirely up to the participants. An Actiwatch will be given to the participants during early pregnancy (12-14 weeks), mid-pregnancy (22-24 weeks), and late pregnancy (29-32 weeks). Instructions will be included on how to wear the watch, with participants advised to wear it on the non-dominant wrist continuously for 7 days, except when swimming or bathing. In addition to the Actiwatch, participants will complete a sleep questionnaire during early pregnancy (12-14 weeks), mid-pregnancy (26-27 weeks), and late pregnancy (35-37 weeks) to subjectively assess their nighttime sleep and napping over the past month. The neurodevelopment of the participants' offspring will be followed up and assessed using the Bayley Scales of Infant and Toddler Development at 6 months, 12 months, 18 months, and 2 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women with a PSQI score greater than 5 at enrollment.
2. Not a habitual napper in the past 3 months (defined as napping 5 or more days per week on average for the past month).

Exclusion Criteria:

Women with severe respiratory or cardiovascular diseases, liver or kidney dysfunction, or malignant tumors.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-19 (Estimated); Primary Completion 2028-08-18 (Estimated); Study Completion 2028-08-18 (Estimated)

PRIMARY OUTCOMES:
Bayley Scales of Infant and Toddler Development score | Children at 24 months
  The Bayley Scales of Infant and Toddler Development (Bayley-III) evaluates five key developmental domains:
  1. Cognitive Development.
  2. Language Development.
  3. Motor Development.
  4. Social-Emotional Development.
  5. Adaptive Behavior.

SECONDARY OUTCOMES:
Ages and Stages Questionnaires (ASQ) score | Children at 12 months
  ASQ typically evaluates the following areas:
  1. Communication.
  2. Gross Motor.
  3. Fine Motor.
  4. Problem Solving.
  5. Personal-Social.
Ages and Stages Questionnaires (ASQ) score | Children at 6 months
  ASQ typically evaluates the following areas:
  1. Communication.
  2. Gross Motor.
  3. Fine Motor.
  4. Problem Solving.
  5. Personal-Social.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Huang, Ph.D., Principal Investigator — Xinhua Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China